CLINICAL TRIAL: NCT02855567
Title: The Role of Acupuncture in Post-Operative Pain Management in Gynecological Patients
Brief Title: Acupuncture for Post-Operative Pain Control for Patients Undergoing Gynecological Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 16-1120
Record Dates: First submitted 2016-07-29; First posted 2016-08-04 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Post-operative Pain; Gynecological Surgery; Acupuncture
Keywords: surgery; acupuncture; gynecology; pain; narcotics
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Acupuncture (Active Comparator): Receives acupuncture during gynecological surgery at 5 known points for pain control. Needles will be placed prior to the start of surgery by an anesthesiologist trained in acupuncture after induction of anesthesia and while the patient is prepped for surgery. They will be in place for 15 minutes.
  Interventions: Device: Acupuncture needles
- Sham acupuncture (Sham Comparator): Receives acupuncture during gynecological surgery at sham points not associated with pain control. Needles will be placed by the gynecologic surgeon who is not trained in acupuncture after induction of anesthesia and prior to the start of the surgery. The needles will be removed immediately after placement.
  Interventions: Device: Acupuncture needles

INTERVENTIONS:
Device: Acupuncture needles — Acupuncture needles (29 and 30 gauge) used to perform the acupuncture

SUMMARY:
This study investigates the role of acupuncture in controlling post-operative pain in patients who have undergone gynecological surgery.

DETAILED DESCRIPTION:
The goal of the study is to investigate acupuncture at the time of gynecological surgery as a way to decrease post-operative pain which would decrease narcotic intake and hospitalization time. To do this, the researchers will recruit non-pregnant patients over the age of 18 who are undergoing laparoscopic surgery for a benign gynecological indication. These patients will be randomized using a computer generated randomization system to receive either acupuncture or sham acupuncture pre-operatively after the induction of anesthesia. The acupuncture points used will be points proven in the literature to be associated with decreasing general pain, pelvic pain and nausea and vomiting. The needles will be placed by a anesthesiologist trained in acupuncture and they will be left in place for 15 minutes while the patient is prepped for the surgery. The sham points will be on the hands and feet and chosen at random by the gynecologic surgeon who is not trained in acupuncture. For both groups, the acupuncture needles will be removed before the first incision of the surgery. All patients will be blinded to their group allocation.

ELIGIBILITY:
Inclusion Criteria:

* female patients
* over the age of 18
* scheduled for laparoscopic gynecological procedures for benign conditions of the uterus, fallopian tubes and/or adnexa

Exclusion Criteria:

* male patients
* pregnancy
* suspected or known malignant disease
* immunocompromised
* known or persistent abuse of medications, drugs or alcohol
* chronic pain for greater than 3 months

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-08-06 (Actual); Primary Completion 2017-12-05 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Ascher-Walsh, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Acupuncture: Received acupuncture during gynecological surgery at 5 known points for pain control. Needles placed prior to the start of surgery by an anesthesiologist trained in acupuncture after induction of anesthesia and while the patient was prepped for surgery. 30-gauge needles were placed for 15 minutes while the patient was positioned and prepped for surgery.
- Sham Acupuncture: Received acupuncture during gynecological surgery at sham points not associated with pain control. The same size needles were placed by the gynecologic surgeon who is not trained in acupuncture after induction of anesthesia and prior to the start of the surgery. The needles were removed immediately after placement.
Period: Overall Study
Arm/Group | Acupuncture | Sham Acupuncture
Started | 54 | 56
Completed | 54 | 56
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 54 | 56 | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.99 (10.84) | 48.58 (12.52) | 45 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 56 | 110
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 35 | 45 | 80
  Unknown or Not Reported | 11 | 6 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 3 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 9 | 14 | 23
  White | 22 | 25 | 47
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 22 | 14 | 36
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 27.17 (6.95) | 27.34 (6.64) | 27.22 (6.70)
Prior abdominal surgery [Count of Participants; unit: Participants] | 21 | 29 | 50
Indication for surgery [Count of Participants; unit: Participants]
  Abnormal Uterine Bleeding (AUB) | 30 | 30 | 60
  Adnexal mass | 2 | 5 | 7
  Bulk | 8 | 6 | 14
  Infertility | 5 | 2 | 7
  Prolapse | 7 | 12 | 19
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Morphine Equivalent Usage While in the Hospital
Description: Effectiveness of intra-operative acupuncture in post-operative pain control as measured by narcotic use in the 24 hours post-operatively. Narcotic use monitored either through hospital records if patient is still admitted to the hospital or over the phone if the patient is discharged home prior to 24 hours post-operative.
Time Frame: Intra-operative and 24 hours post-operatively
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 54 | 56
mg
  Intra-operative | 29.59 (14.42) | 30.82 (12.47)
  24 hours Post-operative | 10.54 (8.33) | 11.74 (10.36)

2. Secondary Outcome: Number of Pain Medication Tablets Used at Home Post-Operatively
Description: Patients kept a log of pain medication use once they were discharged from the hospital for first 7 days post operatively.
Time Frame: 7 days post-operatively
Measure: Median (Inter-Quartile Range); unit: tablets
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 54 | 56
tablets
  oxycodone/acetaminophen tablets | 6 [1.5 to 8] | 4 [0 to 9]
  ibuprofen tablets | 5 [0 to 15.5] | 6.5 [0 to 13.5]

3. Secondary Outcome: Number of Patients Readmitted to the Hospital
Description: Effectiveness of intra-operative acupuncture in post-operative pain control as measured by re-admission to the hospital for pain management.
Time Frame: 2 weeks post-operatively
Measure: Count of Participants; unit: Participants
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 54 | 56
Participants | 0 | 0

4. Secondary Outcome: Pain Score
Description: Pain Score. Patients asked to rate pain score total from 0-10 with higher score indicating more pain
Time Frame: up to 4 hours post operatively
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 54 | 56
score on a scale
  Hour 0 | 2.95 [2.04 to 3.85] | 4.05 [3.19 to 4.90]
  Hour 1 | 4.27 [3.48 to 5.06] | 4.50 [3.67 to 5.33]
  Hour 2 | 3.49 [2.69 to 4.29] | 3.61 [2.80 to 4.42]
  Hour 4 | 3.10 [2.09 to 4.12] | 3.00 [2.00 to 4.00]

5. Secondary Outcome: Pain Score at Home Post-Operatively
Description: Pain Score from 0-10 with higher score indicating more pain
Time Frame: up to 7 days post operatively
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 54 | 56
score on a scale
  Day 1 | 4.62 [3.97 to 5.28] | 5.27 [4.65 to 5.88]
  Day 2 | 4.18 [3.53 to 4.84] | 4.40 [3.78 to 5.02]
  Day 3 | 3.60 [2.94 to 4.25] | 3.73 [3.11 to 4.35]
  Day 4 | 3.03 [2.36 to 3.69] | 3.00 [2.37 to 3.63]
  Day 5 | 2.61 [1.95 to 3.28] | 2.38 [1.75 to 3.00]
  Day 6 | 2.21 [1.55 to 2.88] | 2.06 [1.43 to 2.68]
  Day 7 | 1.93 [1.26 to 2.59] | 1.76 [1.13 to 2.38]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/56
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/56
Other Adverse Events (participants affected / at risk) | 0/54 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-06-19): https://cdn.clinicaltrials.gov/large-docs/67/NCT02855567/Prot_SAP_000.pdf